CLINICAL TRIAL: NCT01045785
Title: Investigation of Platelet Function and Aspirin Resistance in Chronic Dialysis Patient
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jenqwen Huang, Internal Medicine, National Taiwan University Hospital
Other Study IDs: 200912018R
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2009-12

CONDITIONS: End Stage Renal Disease
Keywords: aspirin resistance, platelet function assay, dialysis, end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aspirin responsive: PFA Col/EPI normal
- aspirin resistance: PFA Col/epi showed resistance

SUMMARY:
The purpose of this study is to determine whether aspirin resistance has impact on cardiovascular event in dialysis patient.

DETAILED DESCRIPTION:
Dialysis patient inevitably suffered from uremic bleeding although improvement of dialysis care in the past decades. Physicians used to check bleeding time as a surrogate marker for uremic bleeding. However, bleeding time isn't accurate and as well known, is poorly correlated with clinical bleeding such as surgical bleeding. Platelet function assay (PFA) is a newly developed method to measure platelet aggregation in vitro and is validated in many sorts of platelet disorders. Recently, PFA was also used to evaluate aspirin responsiveness in patients who had taken aspirin. Our study is aim to investigate uremic thrombocytopathy via PFA of dialysis patient in Taiwan. Furthermore, we will study aspirin resistance in dialysis patient.

ELIGIBILITY:
Inclusion Criteria:

* dialysis >3 months
* Hb>10 g/dl & Plt > 10000

Exclusion Criteria:

* using medication which interfere PFA except aspirin
* terminal disease such as malignancy
* active vasculitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dialysis patients which follow-up at least monthly at National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
cardiovascular event, bleeding event,and thrombosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jenqwen Huang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Bilgin AU, Karadogan I, Artac M, Kizilors A, Bligin R, Undar L. Hemodialysis shortens long in vitro closure times as measured by the PFA-100. Med Sci Monit. 2007 Mar;13(3):CR141-5. PMID 17325638
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/17325638